CLINICAL TRIAL: NCT05798078
Title: The Relationship Between Social Anxiety and Anxious Thinking Styles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Utrecht University (Other); University of Osnabrueck (Other)
Responsible Party: Principal Investigator, Marcella Woud, Junior Professor, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 582
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Social Anxiety
Keywords: social anxiety; interpretation bias; cognitive bias modification

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blind as to whether they have been allocated to the active training condition or sham training condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Modification for Interpretation (CBM-I) (Experimental): Participants in this arm complete an initial introductory session of Cognitive Bias Modification for Interpretation (CBM-I) in the lab followed by 6 sessions scheduled to be completed over the subsequent week (1 per day). CBM-I will be administered via an online platform using an individual login account.
  Interventions: Behavioral: Cognitive Bias Modification for Interpretation (CBM-I)
- Sham Training Control Condition (Sham Comparator): Participants in this arm complete an initial introductory session of the sham training control condition in the lab followed by 6 sessions scheduled to be completed over the subsequent week (1 per day). CBM-I will be administered via an online platform using an individual login account.
  Interventions: Behavioral: Sham Training Control Condition

INTERVENTIONS:
Behavioral: Cognitive Bias Modification for Interpretation (CBM-I) — The CBM-I intervention is based on the interpretation training paradigm developed by Mathews and Mackintosh (2000). It comprises a series of training scenarios describing different (mostly everyday) socially-relevant situations, structured so they start ambiguously but always have a positive ending. The positive ending is presented as word fragment, which participants are instructure to complete. In about 25% of trials, participants are further requested to respond to comprehension questions about the scenario presented. Each CBM-I session comprises 45 trials presented in 5 blocks of 9 scenarios.
  Arms: Cognitive Bias Modification for Interpretation (CBM-I)
Behavioral: Sham Training Control Condition — The sham training is in an identical format to the CBM-I training, except that the scenarios are all entirely neutral, with no reference to social situations and no emotional ambiguity.
  Arms: Sham Training Control Condition

SUMMARY:
This study aims to investigate whether reductions in negative interpretation biases, induced via an experimental manipulation (Cognitive Bias Modification for Interpretation; CBM-I), lead to reductions in symptoms of social anxiety amongst individuals experiencing high levels of social anxiety. The study further aims to investigate the relationship between multifaceted measures of interpretation bias, psychopathological symptoms, neurophysiological indices, behavioral indices of stress reactivity, and SAD symptoms.

To achieve these aims a sample of individuals experiencing high levels of social anxiety will be recruited. After completing multi-faceted measures of interpretation bias, including neurophysiological indices, participants will be randomized to complete an online one-week daily CBM-I or sham training control condition training schedule. Following the one week training, individuals will return to the lab to complete further multi-faceted measures of interpretation bias and social anxiety symptoms. One week after this (i.e. 2 weeks post-basline), participants will complete a final set of symptom and bias measures online.

ELIGIBILITY:
Inclusion Criteria:

* Provides informed consent
* Sufficient German language skills to complete the experimental tasks and questionnaires
* Aged between 18 and 65 years
* Scoring ≥ 52 on the SPAI-G (Turner et al., 1989; Fydrich, 2016), indicating elevated levels of social anxiety
* Lives within reasonable travelling distance of the research centre

Exclusion Criteria:

* Current psychotherapeutic treatment or psychotherapeutic treatment completed within the last 6 months prior to study enrolment.
* Current substance misuse or dependency (apart from Nicotine)
* Acute suicidality or self-harm
* Symptoms of a psychotic or bipolar disorder
* Presence of a somatic condition that could systematically affect cortisol levels (in particular: Pregnancy and lactation, adrenal dysfunction, thyroid dysfunction, pituitary dysfunction)
* Presence of a somatic condition that could systematically affect brain physiology (current or anamnestic neurological disorders, in particular: anamnestic traumatic brain injury, epilepsy, multiple sclerosis, brain tumors)
* Presence of a somatic condition that could systematically affect peripheral physiological measures (in particular: cardiovascular diseases (e.g., cardiac arrhythmias, circulatory diseases [e.g., hypertension]))
* Sensitivity or alteration of skin surface providing contraindication for EEG or periphysiological measures (in particular: baldness, dreadlocks, open wounds on the head or facial surface, skin conditions that cause particular sensitivity to gels and creams)
* Intake of psychotropic medication that cannot be interrupted during study duration or change in psychotropic medication within the 8 weeks before starting the study (except: antidepressants in unaltered dosage)
* Left handedness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline to follow-up (2 weeks post-baseline) in score on the Liebowitz Social Anxiety Scale, Self-Report (LSAS-SR) | Baseline, Follow-up (2 weeks post-baseline)
  A 24-item self-report scale assessing social anxiety symptoms over the past 7 days (Consbruch, Stangier & Heidenreich, 2016; Liebowitz, 1987). Possible scores range from 0 (minimum) to 144 (maximum), with higher scores reflecting higher levels of social anxiety (i.e. worse outcomes). The primary outcome measure is change in score on the LSAS-SR from baseline to follow-up.

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale, Self-Report (LSAS-SR) | Post-training (1 week post-baseline)
  A 24-item self-report scale assessing social anxiety symptoms over the past 7 days (Consbruch, Stangier & Heidenreich, 2016; Liebowitz, 1987). Possible scores range from 0 (minimum) to 144 (maximum), with higher scores reflecting higher levels of social anxiety (i.e. worse outcomes).
Social Phobia and Anxiety Inventory, German version (SPAI-G) | Screening, Baseline, Post-training (1 week post-baseline), Follow-up (2 weeks post-baseline)
  A 22-item self-report scale used for screening different levels of social anxiety (Turner et al., 1989; Fydrich, 2016). Possible scores range from 0 (minimum) to 132 (maximum), with higher scores reflecting higher levels of social anxiety (i.e. worse outcomes).
Depression, Anxiety, and Stress Scale-21 (DASS) | Baseline, Post-training (1 week post-baseline), Follow-up (2 weeks post-baseline)
  A 21-item self-report questionnaire assessing symptoms of depression, stress and anxiety (7 items per subscale) over the past week (Lovibond & Lovibond, 1995; Nilges & Essau, 2015). Possible scores on each subscale range from 0 (minimum) to 21 (maximum), with higher scores reflecting higher levels of symptoms (i.e. worse outcomes).
Brief Fear of Negative Evaluation Scale (BFNE) | Baseline, Post-training (1 week post-baseline), Follow-up (2 weeks post-baseline)
  A 12-item self-report scale used to assess fear of being negatively evaluated by others in social situations (Leary, 1983; Reichenberger, Schwarz, König, Wilhelm, .. & Blechert, 2016). Possible scores range from 12 (minimum) to 60 (maximum), with higher scores reflecting higher levels of fear (i.e. worse outcomes).
Encoding Recognition Task (ERT) | Baseline, After last intervention session (~6 days post-baseline), Post-training (1 week post-baseline), Follow-up (2 weeks post-baseline)
  The ERT is a 10-item computerized measure of interpretation bias (Salemink & van den Hout, 2010). Four versions are used, applied in a counterbalanced order across participants.
Scenario Rating Task (SRT) | Baseline, Post-training (1 week post-baseline)
  The SRT is used to assess interpretation biases and their neurophysiological correlates via EEG (N400). Participants read ambiguous scenarios (i.e., sentence stems) that are completed by either congruent or incongruent endings, and have to rate how well the endings complete the sentence stems. Participants will be presented with a total of 96 trials, 48 of which are neutral and 48 of which are social anxiety-related. In addition to behavioural responses, the N400 amplitude will be measured via EEG in the 300-450 ms time window post-stimulus onset (i.e., the target word, e.g., Feng et al., 2019; Moser et al., 2008).
Anagram Task | Post-training (1 week post-baseline)
  The Anagram task is used to investigate stress reactivity towards social-evaluative threats in performance situations (Van Bockstaele et al., 2020). During the Anagram Task, heart rate, heart rate variability, and corrugator activity will be recorded. The state mood ratings (listed below) are used to measure mood response to the task.
Salivary cortisol | Baseline, Post-training (1 week post-baseline)
  Salivary concentrations of cortisol will be collected during both lab assessments. During the first lab assessment, it will be collected once at baseline prior to the administration of the questionnaires. During the second lab assessment, it will be collected four times, at baseline prior to the administration of the questionnaires, pre-Anagram Task, post-Anagram task, post-Anagram task+25 min.
Salivary alpha-amylase | Baseline, Post-training (1 week post-baseline)
  Salivary concentrations alpha-amylase will be collected during both lab assessments. During the first lab assessment, it will be collected once at baseline prior to the administration of the questionnaires. During the second lab assessment, it will be collected four times, at baseline prior to the administration of the questionnaires, pre-Anagram Task, post-Anagram task, post-Anagram task+25 min.
Frontal Asymmetry | Baseline, Post-training (1 week post-baseline)
  Following Moscovitch et al. (2011), resting frontal alpha asymmetry will be recorded using EEG during an 8-minute resting period (in alternating 1-min eyes-open/eyes-closed segments) at both pre- and post-training. In addition, frontal assymetry will be recorded during the SRT, i.e., when presenting the ambiguous stems.

OTHER OUTCOMES:
Expectancy Questionnaire (EQ) | Baseline
  Expectancy effects will be assessed prior to training using the three expectancy items from the Credibility and Expectancy Questionnaire (Borkovec & Mathews, 1988). A total score is made by standardizing (z-transforming) the three items and adding the z-transformed scores together (i.e. no minimum or maximum scores). Higher scores indicate higher expectancy of improvement.
Feedback Questionnaire | Follow-up (2 weeks post-baseline)
  A questionnaire asking for feedback about the CBM/Sham intervention will be used, adapted from Woud et al. (2021). Each individual item is interpreted separately (i.e. no sum score is created).
Negative Effects Questionnaire (NEQ) | Follow-up (2 weeks post-baseline)
  The short (20-item) version of the Negative Effects Questionnaire (Rozental et al., 2019) will be used to assess potential negative effects and adverse events linked to the study. The scale will be adapted for the purpose of the study with terms like 'therapy' and 'therapist' changed to e.g. 'study' and 'researchers' (as per Blackwell et al., 2022). The number of reported negative effects for each category are summed for reporting purposes.
State affect | Baseline, Post-training (1 week post-training)
  State affect will be measured repeatedly throughout the assessment sessions (i.e., at baseline, pre-stressor, post-stressor, during and after the recovery phase) using a 7-item scale developed by Becker et al. (2016). This scale includes the following items: "I feel… tense / sad / anxious / confident / relaxed / happy / relieved", with each item being judged via a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marcella L Woud, PhD, Principal Investigator — Ruhr University of Bochum
Locations (1):
- Mental Health Research and Treatment Center, Ruhr University of Bochum, Bochum, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on publication via a suitable repository such as the Open Science Framework, and will be made available to reviewers at the time of submission (or publically with a pre-print version of the manuscript). Data made available will be the research data reported in the publication, withthe exception of any data that could compromise participant anonymity.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Supporting information will be made available on publication via a suitable repository such as the Open Science Framework, and will be made available to reviewers at the time of submission (or publically with a pre-print version of the manuscript).
URL: https://osf.io/e254p/